CLINICAL TRIAL: NCT04167306
Title: A Randomized, Double-blind, Placebo-controlled Multicenter Trial on the Efficacy of Varenicline and Bupropion in Combination and Alone, for Treatment of Alcohol Use Disorder
Brief Title: Varenicline and Bupropion for Alcohol Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COMB-BO8; 2018-000048-24 (EudraCT Number)
Record Dates: First submitted 2019-09-30; First posted 2019-11-18 (Actual); Results first posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2023-12

CONDITIONS: Alcohol Use Disorder; Alcoholism; Alcohol Dependence
MeSH Terms: conditions — Alcoholism | interventions — Varenicline; Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Appointed manufacturer produces, packs and labels the IMPs in two separate IMP kits and uses a blinding procedure accordance with internal standard operating procedure. IMP 1 and IMP 2, will have an unique Randomization Number generated randomly. For each randomization number, a sealed emergency code envelope will follow the shipment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1) Varenicline + Bupropion (Experimental): Investigational medicinal product (IMP) 1: Varenicline 0.5 mg and 1.0 mg and Investigational medicinal product (IMP) 2: Bupropion SR 150 mg
  Interventions: Drug: Varenicline Tartrate 1 mg b.i.d; Drug: Bupropion Hydrochloride 150 mg b.i.d
- 2) Varenicline + Placebo for Bupropion (Experimental): Investigational medicinal product (IMP) 1: Varenicline 0.5 mg and 1.0 mg and Placebo capsule for IMP 2 (bupropion)
  Interventions: Drug: Varenicline Tartrate 1 mg b.i.d; Other: Placebo for bupropion
- 3) Bupropion + Placebo for Varenicline (Experimental): Investigational medicinal product (IMP) 2: Bupropion SR 150 mg and Placebo capsule for IMP 1 (varenicline)
  Interventions: Drug: Bupropion Hydrochloride 150 mg b.i.d; Other: Placebo for varenicline
- 4) Placebo for Varenicline + Placebo for Bupropion (Placebo Comparator): Placebo capsule for IMP 1 (varenicline) and Placebo capsule for IMP 2 (bupropion)
  Interventions: Other: Placebo for varenicline; Other: Placebo for bupropion

INTERVENTIONS:
Drug: Varenicline Tartrate 1 mg b.i.d — Capsules for oral use
  Other Names: Champix
  Arms: 1) Varenicline + Bupropion; 2) Varenicline + Placebo for Bupropion
Drug: Bupropion Hydrochloride 150 mg b.i.d — Capsules for oral use
  Other Names: Bupropion Sandoz
  Arms: 1) Varenicline + Bupropion; 3) Bupropion + Placebo for Varenicline
Other: Placebo for varenicline — Capsules for oral use
  Arms: 3) Bupropion + Placebo for Varenicline; 4) Placebo for Varenicline + Placebo for Bupropion
Other: Placebo for bupropion — Capsules for oral use
  Arms: 2) Varenicline + Placebo for Bupropion; 4) Placebo for Varenicline + Placebo for Bupropion

SUMMARY:
The COMB study is a randomized double-blind placebo-controlled multicenter trial in Sweden on the efficacy of varenicline and bupropion, in combination and alone, for treatment of alcohol use disorder (AUD).

Study design overview: A 13-weeks (91 days) multicenter clinical trial with four parallel groups. 95 subjects per treatment arm will be randomized into the study. 380 subjects with AUD will be randomized in total.

DETAILED DESCRIPTION:
Varenicline (Champix®) and bupropion (Zyban®, patent time expired) are approved and marketed in Europe and US for smoking cessation in nicotine use disorder, and for treatment of major depression (bupropion). There is clinical evidence of an additive effect of the drug combination of varenicline and bupropion on smoking cessation. Varenicline has been shown in two RCTs to reduce also alcohol intake in subjects with AUD. It is hypothesized that bupropion will enhance the effect of varenicline and that the combined effect size will be greater than that of approved therapies for AUD. As efficacy endpoint, the trial uses the alcohol specific biomarker for alcohol intake, phosphatidylethanol in blood (B-PEth). Outcome will also be measured by self-reported alcohol consumption, the standard effect measure in AUD trials.This will be the first trial using the biomarker B-PEth as primary outcome variable. The use of a specific objective marker is expected to increase chances for detecting treatment effects.

Development phase: II Number of randomized subjects: 380 subjects with AUD. 95 subjects per treatment arm will be randomized into the study.

Number of sites: Approximately 5 study sites in Sweden

Investigational medicinal products, dosages and administration:

There will be two separate study kits for IMP 1 and IMP 2

Investigational medicinal product 1 (IMP1): Varenicline 1 mg x 2 p.o. daily. The pharmaceutical formulation will be encapsulated tablets for oral use. Varenicline will be escalated from 0.5 to 2 mg daily during the first week.

Investigational medicinal product 2 (IMP 2): Bupropion SR 150 mg x 2 p.o. daily. The pharmaceutical formulation will be encapsulated sustained release (SR) tablets for oral use. Bupropion will be escalated from 150 to 300 mg daily during the first week.

IMP 1 and IMP 2 are distributed at 7 occasions: Day 0, Day 7, Day 21, Day 35, Day 49, Day 63 and Day 77. The doses and route of administration for varenicline and bupropion are those approved and recommended as oral formulations for smoking cessation.

The trial comprises 9 study visits over 91 days: Screening visit,Day 0, Day 7, Day 21, Day 35, Day 49, Day 63, Day 77 and Day 91. Randomization is carried out according to block randomization and eligible subjects are randomized to one of the below described intervention arms.

The study will be performed in accordance with the study protocol, with the latest version of the Declaration of Helsinki, in accordance with GCP principles (ICH-GCP E6-R2), and applicable regulatory requirements in Sweden . The study is approved by competent authority (the Swedish Medical Product Agency) and the Etics committee. The trial is monitored by an independent monitor according to GCP principles.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Blood alcohol level below <0.1‰ (0.1 g/L) at signing informed consent
3. 25-70 years of age at screening
4. Moderate and severe AUD according to DSM-V (meeting ≥4 out of 11 criteria)
5. B-PEth levels of ≥0.5 µmol/L at screening visit (visit 1)
6. Continuous high alcohol consumption over the last 3 months prior to screening as defined by at least 2 HDD per week on a typical week
7. Available phone number for contact
8. Ability to speak and write in Swedish

Exclusion Criteria:

1. Total abstinence between screening and randomization visit
2. Treatment of alcohol withdrawal within 30 days of study initiation
3. Pharmacological treatment within 3 months of study initiation and during the study period that may affect alcohol consumption, including but not exclusive to, varenicline, bupropion, disulfiram, acamprosate, naltrexone, nalmefene, baclofen, topiramate, ondansetron, mirtazapine, methylphenidate, dexamphetamine, atomoxetine, pregabalin, buprenorphine and methadone
4. Non-pharmacological treatment within 3 months of study initiation and during the study period that may affect alcohol consumption
5. Current continuous use of antidepressants, opioid analgesics, benzodiazepines, zopiclone, zolpidem, hydroxyzine, alimemazine, propiomazine, or other sedatives. (The sporadic use of these compounds is accepted.)
6. Any concurrent medication that may affect the results of the trial or is considered to compromise the safety of the participants in the trial. (See SmPCs for possible interactions.)
7. Laboratory hepatic values of >3 times the upper limit of the normal range, creatinine clearance <30 ml/min, or other clinically significant abnormalities in the screening laboratory values
8. Blood pressure ≥180/110 at screening
9. Pregnancy, breast-feeding and for premenopausal women, not using one of the contraceptive methods oral contraceptive, intrauterine contraceptive device (copper or hormonal) or subcutaneous inplant.
10. Diabetes mellitus type 1 and diabetes mellitus type 2 in need of insulin treatment
11. Any current psychiatric or somatic disorder or condition that may affect assessments or compromise participant's safety during the trial
12. ASRS- v1.1, part A score ≥4 in the marked cut-off section
13. MADRS score ≥ 20
14. Current depression that is not mild (mild depression is accepted)
15. Suicidality
16. Current illicit drug use based on urine-toxicity test and DUDIT
17. History of delirium tremens or abstinence-induced seizures within 5 years of study initiation
18. Epilepsy or seizures other than alcohol-induced, lifetime
19. Severe sleep disturbances
20. Need of alcohol detoxification
21. Living conditions not appropriate to fulfil study requirements
22. Use of herbal drugs/tea and supplementations possibly affecting outcome or safety
23. Previous randomization in this trial or participation in another trial within 3 months of enrollment into this trial.
24. Additional factors that render the participant unable to complete the study, as judged by the investigator

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bo Söderpalm, Prof, MD, Principal Investigator — Sahlgrenska University Hospital, Västra Götaland
Locations (4):
- Sweden (4):
  - Beroendecentrum Malmö, Malmo, Region Skåne
  - Linköping University Hospital, Linköping, Region Östergötland
  - Stockholm Centre for Dependency Disorders,, Stockholm, Stockholms Läns Sjukvårdområde
  - Beroendekliniken, Sahlgrenska University Hospital, Västra Götalandsregionen, Gothenburg

REFERENCES:
- [Derived] Soderpalm B, Lido H, Franck J, Hakansson A, Lindqvist D, Heilig M, Guterstam J, Samuelson M, Askerup B, Wallmark-Nilsson C, de Bejczy A. Efficacy and safety of varenicline and bupropion, in combination and alone, for alcohol use disorder: a randomized, double-blind, placebo-controlled multicentre trial. Lancet Reg Health Eur. 2025 May 13;54:101310. doi: 10.1016/j.lanepe.2025.101310. eCollection 2025 Jul. PMID 40487775
- [Derived] de Bejczy A, Lido H, Soderpalm B. A randomized, double-blind, placebo-controlled, multicentre trial on the efficacy of varenicline and bupropion in combination and alone for treatment of alcohol use disorder: Protocol for the COMB study. PLoS One. 2024 Jan 11;19(1):e0296118. doi: 10.1371/journal.pone.0296118. eCollection 2024. PMID 38206930

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 2) Varenicline + Placebo for Bupropion | 1) Varenicline + Bupropion | 3) Bupropion + Placebo for Varenicline | 4) Placebo for Varenicline + Placebo for Bupropion
Started | 97 | 101 | 93 | 97
Correct Randomized , Received IMP (correctly randomized subjects that commenced study drug) | 96 | 100 | 91 | 97
Completed | 76 | 73 | 67 | 81
Not Completed | 21 | 28 | 26 | 16
Not completed — Lost to Follow-up | 2 | 2 | 5 | 5
Not completed — Adverse Event | 13 | 14 | 5 | 4
Not completed — Withdrawal by Subject | 4 | 6 | 8 | 3
Not completed — covid | 1 | 1 | 2 | 1
Not completed — concomitant medication | 0 | 0 | 0 | 1
Not completed — Alcohol treatment | 0 | 4 | 3 | 2
Not completed — non-compliance | 0 | 0 | 1 | 0
Not completed — incorrectly randomized or did not commence study drug | 1 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population mITT (modified Intention to Treat) defined as subjects that have taken at least one dose of study drug and documented at least one data entry
Groups:
- Total: Total of all reporting groups
Arm/Group | 1) Varenicline + Bupropion | 2) Varenicline + Placebo for Bupropion | 3) Bupropion + Placebo for Varenicline | 4) Placebo for Varenicline + Placebo for Bupropion | Total
Number analyzed (Participants) | 100 | 96 | 91 | 97 | 384
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (8.3) | 56 (9.7) | 56 (9.2) | 56 (9.9) | 56 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 27 | 18 | 34 | 107
  Male | 72 | 69 | 73 | 63 | 277
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Phosphatidylethanol (B-PEth) [Mean (Standard Deviation); unit: mikromol/L] | 1.2 (0.66) | 1.2 (0.76) | 1.3 (0.62) | 1.2 (0.55) | 1.2 (0.65)
Heavy Drinking Days (HDD) [Mean (Standard Deviation); unit: proportion] | 0.72 (0.30) | 0.76 (0.25) | 0.75 (0.26) | 0.74 (0.28) | 0.74 (0.27)
Age at Alcohol debut [Mean (Standard Deviation); unit: years] | 15 (3.0) | 15 (4.1) | 15 (2.7) | 16 (5.3) | 16 (3.9)
Heredity for alcohol problems [Count of Participants; unit: Participants] | 25 | 15 | 17 | 16 | 73

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Consumption as Measured by Phosphatidylethanol (PEth) in Blood
Description: B-PEth: Objective marker for alcohol consumption measured in blood, measured at every study visit. Analysed as mean reduction of PEth per treatment arm, mITT.
Time Frame: PEth is calculated as the mean value over the active steady state period (Day 21-Day77) compared to baseline (=screening visit value)
Population: modified ITT (mITT), defined as participants taken at least one dose of study drug and documented at least one data entry
Measure: Mean (Standard Error); unit: mikromol/litre
Arm/Group | 2) Varenicline + Placebo for Bupropion | 1) Varenicline + Bupropion | 3) Bupropion + Placebo for Varenicline | 4) Placebo for Varenicline + Placebo for Bupropion
Number analyzed (Participants) | 96 | 100 | 91 | 97
mikromol/litre | -0.406 (0.057) | -0.417 (0.041) | -0.315 (0.054) | 0.250 (0.044)

2. Primary Outcome: Alcohol Consumption as Measured by Heavy Drinking Days (HDD)
Description: HDD is obtained by the time Line Follow Back procedure, defined as ≥70 grams for men and ≥56 grams for women according to FDA's guidelines. Analysed as mean reduction in HDD share per treatment arm, for mITT
Time Frame: Number of HDD by 14 days is defined as a mean over the 8-week steady state active treatment period (Day 21-Day77) . ( D21-D77)/4 in order to get a 14 day-period measurment.
Population: modified ITT (mITT), defined as subjects taken at least one dose of study drug and documented at least one data entry.
Measure: Mean (Standard Error); unit: proportion
Arm/Group | 2) Varenicline + Placebo for Bupropion | 1) Varenicline + Bupropion | 3) Bupropion + Placebo for Varenicline | 4) Placebo for Varenicline + Placebo for Bupropion
Number analyzed (Participants) | 96 | 100 | 91 | 97
proportion | -0.322 (0.028) | -0.314 (0.031) | -0.298 (0.035) | -0.217 (0.031)

3. Secondary Outcome: CDT
Description: The indirect alcohol marker carbohydrate deficient transferrin
Time Frame: CDT is calculated as the mean value over the active steady state period (Day 21-Day77) compared to baseline (=screening visit value)
Reporting Status: Not Posted

4. Secondary Outcome: GGT
Description: The indirect alcohol marker gamma glutamyl transferase
Time Frame: GGT calculated as the mean value over the active steady state period (Day 21-Day77) compared to baseline (=screening visit value)
Reporting Status: Not Posted

5. Secondary Outcome: Self-reported Alcohol Consumption Measured by Time-lime-follow-back
Description: Mean grams of alcohol per day
  * Number of drinking days
  * Number of drinks per drinking days
  * Number of abstaining days
Time Frame: as for outcome 3
Reporting Status: Not Posted

6. Secondary Outcome: Alcohol Use Identification Test
Description: Total score of Alcohol Use Identification Test
Time Frame: Mean difference between total score obtained at baseline and visit 1
Reporting Status: Not Posted

7. Secondary Outcome: Self-reported Alcohol Craving
Description: Alcohol craving as measured by a Visual Analogue Scale (VAS)
Time Frame: Scale range: 0-100 mm. Minimum value: 0 = No craving. Maxumum value: 100 Maximum= Very strong craving. Craving is calculated as the mean value over the active steady state period (Day 21-Day77) compared to baseline (=screening visit value)
Reporting Status: Not Posted

8. Secondary Outcome: Nicotine Use
Description: Nicotine use measured by the nicotine saliva marker cotinine in saliva
Time Frame: 77 day-interval. Mean difference between cotinine concentration assessed at Day o and Day 77
Reporting Status: Not Posted

9. Secondary Outcome: The Temporal Experience of Pleasure Scale (TEPS)
Description: A 17-item scale with anticipatory and consummatory components of the experience of pleasure. The scale is used as a proxy to assess a hypodopaminergic state. Worse Outcome: A lower score indicates low experience of pleasure (=proxy for hypodopaminergic state). Better outcome:A high score indicates high experience of pleasure.
Time Frame: 77 day-interval. Mean difference between total scale score assessed at Day 0 and Day 77
Reporting Status: Not Posted

10. Secondary Outcome: The Continous Performance Test + Activity Test
Description: A neuropsychiatric tool addressing inattention, impulsivity and activity
Time Frame: 77 day-interval. Mean difference between outcome measure assessed at Day o and Day 7.
Reporting Status: Not Posted

11. Secondary Outcome: Plasma Concentration of Varenicline (ng/ml)
Description: Mean concentration of values obtained at visit 4 and visit 6
Time Frame: 14 day-interval. Obtained twice, at Day 21 and Day 49 during IMP steady state. Correlation between plasma concentration of varenicline and above described outcome measures
Reporting Status: Not Posted

12. Secondary Outcome: Plasma Concentration of Bupropion (ng/ml)
Description: Mean concentration of values obtained at visit 4 and visit 6
Time Frame: 14 day-interval. Obtained twice, at Day 21 and Day 49 during IMP steady state. Correlation between plasma concentration of bupropion and above described outcome measures
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: from inclusion (at informed consent) until last Follow-up at 30 days after study drug termination
Description: safety population is equal to mITT population, subjects receiving at least one dose of study drug, N=384
Arm/Group | 2) Varenicline + Placebo for Bupropion | 1) Varenicline + Bupropion | 3) Bupropion + Placebo for Varenicline | 4) Placebo for Varenicline + Placebo for Bupropion
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/100 | 0/91 | 0/97
Serious Adverse Events (participants affected / at risk) | 3/96 | 2/100 | 3/91 | 3/97
Other Adverse Events (participants affected / at risk) | 92/96 | 98/101 | 82/91 | 84/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2) Varenicline + Placebo for Bupropion (N=96) | 1) Varenicline + Bupropion (N=100) | 3) Bupropion + Placebo for Varenicline (N=91) | 4) Placebo for Varenicline + Placebo for Bupropion (N=97)
heart failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
pulmonary embolism (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
malignt melanoema of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
tachycardia irregular (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
calculus of gallbladder with acute cholecystitis, with obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2) Varenicline + Placebo for Bupropion (N=96) | 1) Varenicline + Bupropion (N=101) | 3) Bupropion + Placebo for Varenicline (N=91) | 4) Placebo for Varenicline + Placebo for Bupropion (N=97)
anxiety (Psychiatric disorders) | 9 (9) | 9 (9) | 7 (7) | 2 (2)
arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 7 (7) | 7 (7)
back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1) | 5 (5) | 7 (7)
increased blood pressure (Cardiac disorders) | 6 (6) | 6 (6) | 4 (4) | 7 (7)
cough (Infections and infestations) | 8 (8) | 7 (7) | 6 (6) | 7 (7)
depressed mood (Psychiatric disorders) | 15 (16) | 13 (16) | 13 (16) | 16 (16)
dizziness (Nervous system disorders) | 14 (14) | 5 (5) | 15 (15) | 1 (1)
diarrhea (Gastrointestinal disorders) | 8 (8) | 3 (3) | 4 (4) | 8 (8)
dry mouth (Nervous system disorders) | 5 (5) | 11 (11) | 6 (6) | 4 (4)
fatigue (Psychiatric disorders) | 23 (23) | 9 (9) | 12 (12) | 11 (11)
headache (Nervous system disorders) | 35 (35) | 39 (39) | 27 (27) | 40 (40)
increased hepaic enzymes (Gastrointestinal disorders) | 8 (8) | 3 (3) | 7 (7) | 11 (11)
insomnia (Psychiatric disorders) | 16 (16) | 18 (18) | 15 (15) | 10 (10)
nasopharyngitis (Infections and infestations) | 26 (26) | 27 (27) | 18 (18) | 23 (23)
nausea (Gastrointestinal disorders) | 61 (61) | 38 (38) | 12 (12) | 11 (11)
pyrexia (Infections and infestations) | 3 (3) | 6 (6) | 8 (8) | 3 (3)
sleep disorder (Psychiatric disorders) | 4 (4) | 9 (9) | 2 (2) | 6 (6)
vertigo (Nervous system disorders) | 6 (6) | 8 (8) | 5 (5) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-16): https://cdn.clinicaltrials.gov/large-docs/06/NCT04167306/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-13): https://cdn.clinicaltrials.gov/large-docs/06/NCT04167306/SAP_001.pdf